CLINICAL TRIAL: NCT00215969
Title: Prospective Study of Hypercoagulation in Pregnant Women
Brief Title: Prospective Study in Pregnant Women With Hypercoagulopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Department of Clinical Trials, Denmark (Other Government); Loyola University (Other)
Other Study IDs: PR0104
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2005-09

CONDITIONS: Pre-Eclampsia; Eclampsia
Keywords: Pre-eclampsia; Pregnancy; Hypercoagulation; Screening; Cardiovascular complications
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; Thrombophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Pre-eclampsia is one of the most common causes of maternal and fetal morbidity and mortality. The aim of this study is to identify pregnant women at risk for pre-eclampsia or other cardiovascular complications at a very early state of the disease, and thereby improve the current method of screening.

DETAILED DESCRIPTION:
600 pregnant women will be included in the project and followed in a standardized manner during their pregnancy. On a regular basis blood- and urine samples will be taken throughout their pregnancy and until 1 month after delivery and analyzed for a large variety of coagulation factors in order to identify factors that might predict an increased risk of developing pre-eclampsia and/or cardiovascular events. In addition a DNA-sample is taken if consented in order to evaluate genetic factors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending the midwife at Hilleroed Hospital, Frederiksborg County, Denmark.

Exclusion Criteria:

* Mental disease.
* Problems understanding or reading Danish.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-01; Study Completion 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Anita S Andersen, MD, Principal Investigator
Locations (2):
- Denmark (2):
  - Department of Gynaecology and Obstetrics, Hilleroed Hospital, Hilleroed, Frederiksborg County
  - Department of Gynaecology and Obstetrics, Hilleroed, Frederiksborg